CLINICAL TRIAL: NCT00246987
Title: A Phase 3, Randomized, Double-blind, Placebo Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of BMS-298585 as Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: A Trial to Evaluate BMS-298585 as Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV168-018
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — muraglitazar

INTERVENTIONS:
Drug: Muraglitazar

SUMMARY:
To determine the effect on glycemic control and lipid parameters of the 2.5 and 5 mg. doses of BMS-298585 in drug naive subjects with Type 2 diabetes as an adjunct to diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 diabetes
* Drug Naive
* HbA1c >= 7.0% and <= 10.0%
* Body Mass Index <= 41 kg/m2
* Serum TG <= 600 mg/dL

Exclusion Criteria:

* Symptomatic Type 2 diabetes
* History of bladder cancer
* History of Myocardial Infarction (MI), coronary angioplasty or bypass grafts, valvular disease or repair, unstable angina pectoris, Transient Ischemic Attach (TIA), or Cerebrovascular Accident (CVA) within 6 months, congestive heart failure (NYHA Class II and IV), uncontrolled hypertension, history of renal disease, peripheral vascular disease (PVD), pulmonary disease, gastrointestinal disease, active liver disease or endocrine disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341
Dates: Start 2003-06; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to Week 24

SECONDARY OUTCOMES:
Changes achieved from baseline in FPG after 24 weeks. Changes achieved from baseline in 3 hour post-prandial AUC for glucose and insulin levels after 24 weeks vs. placebo.

CONTACTS AND LOCATIONS:
Locations (130):
- United States (82):
  - Local Institution, Anniston, Alabama
  - Local Institution, Birmingham, Alabama
  - Local Institution, Haleyville, Alabama
  - Local Institution, Hoover, Alabama
  - Local Institution, Fayetteville, Arizona
  - Local Institution, Hot Springs, Arizona
  - Local Institution, Mesa, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Tulsa, Arizona
  - Local Institution, Concord, California
  - Local Institution, Fountain Valley, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Gatos, California
  - Local Institution, Raleigh, California
  - Local Institution, Roseville, California
  - Local Institution, San Diego, California
  - Local Institution, Spring Valley, California
  - Local Institution, Tustin, California
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Golden, Colorado
  - Local Institution, Littleton, Colorado
  - Local Institution, New Britain, Connecticut
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Brandon, Florida
  - Local Institution, Chipley, Florida
  - Local Institution, Coral Gables, Florida
  - Local Institution, Kissimmee, Florida
  - Local Institution, Longwood, Florida
  - Local Institution, Melbourne, Florida
  - Local Institution, New Port Richie, Florida
  - Local Institution, Ocala, Florida
  - Local Institution, Pinellas Park, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Overland Park, Kansas
  - Local Institution, Shawnee Mission, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Madisonville, Kentucky
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Gulfport, Mississippi
  - Local Institution, Saint Peters, Mississippi
  - Local Institution, Chesterfield, Missouri
  - Local Institution, Kansas City, Missouri
  - Local Institution, Springfield, Missouri
  - Local Institution, Elizabeth, New Jersey
  - Local Institution, Toms River, New Jersey
  - Local Institution, Endwell, New York
  - Local Institution, West Seneca, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, High Point, North Carolina
  - Local Institution, Morehead City, North Carolina
  - Local Institution, Salisbury, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Franklin, Ohio
  - Local Institution, Newark, Ohio
  - Local Institution, Zanesville, Ohio
  - Local Institution, Eugene, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Reading, Pennsylvania
  - Local Institution, Warminster, Pennsylvania
  - Local Institution, East Providence, Rhode Island
  - Local Institution, Johnston, Rhode Island
  - Local Institution, Providence, Rhode Island
  - Local Institution, Anderson, South Carolina
  - Local Institution, Greer, South Carolina
  - Local Institution, Mt. Pleasant, South Carolina
  - Local Institution, Knoxville, Tennessee
  - Local Institution, Memphis, Tennessee
  - Local Institution, Fort Worth, Texas
  - Local Institution, Lubbock, Texas
  - Local Institution, San Angelo, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Richmond, Virginia
  - Local Institution, Virginia Beach, Virginia
  - Local Institution, Edmonds, Washington
  - Local Institution, Federal Way, Washington
  - Local Institution, Olympia, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Vancouver, Washington
  - Local Institution, Milwaukee, Wisconsin
- Australia (9):
  - Local Institution, Canberra, New South Wales
  - Local Institution, Sydney, New South Wales
  - Local Institution, Wollongong, New South Wales
  - Local Institution, Kippa-Ring, Queensland
  - Local Institution, Meadowbrook, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Woodville, South Australia
  - Local Institution, Launceston, Tasmania
  - Tasmania, Melbourne, Victoria
- Canada (25):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Coquitlam, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Manuels, Newfoundland and Labrador
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Markham, Ontario
  - Local Institution, Oakville, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Thornhill, Ontario
  - Local Institution, Thunder Bay, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Chicoutimi, Quebec
  - Local Institution, Drummondville, Quebec
  - Local Institution, Granby, Quebec
  - Local Institution, Laval, Quebec
  - Local Institution, Longueuil, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Pointe-Claire, Quebec
  - Local Institution, Saint-Lambert, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Regina, Saskatchewan
  - Local Institution, Saskatoon, Saskatchewan
- Mexico (4):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Durango, Durango
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Cuernavaca, Morelos
- Poland (5):
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Mroków
  - Local Institution, Warsaw
  - Local Institution, Zabrze
- Puerto Rico (3):
  - Local Institution, Añasco
  - Local Institution, Ponce
  - Local Institution, Rio Pieoras
- Taiwan (2):
  - Local Institution, Changhua
  - Local Institution, Taichung